CLINICAL TRIAL: NCT01643213
Title: Randomized Study of Failed SCS Trials Comparing Outcomes Using the Observational Mechanical Gateway (OMG) Connector
Acronym: RESCUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A7006; A7006 (Other: Boston Scientific)
Record Dates: First submitted 2012-07-11; First posted 2012-07-18 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BSC approved SCS Trial Therapy w/ OMG (Experimental): Precision Plus SCS Trial Therapy w/ OMG. Spinal cord stimulation (SCS) trial therapy activated using FDA-approved BSC SCS trial systems with the Observational Mechanical Gateway(OMG) to connect to non-BSC lead(s)
  Interventions: Device: BSC approved SCS Trial Therapy w/ OMG
- Non Boston Scientific SCS Trial Therapy (Active Comparator): Non Boston Scientific SCS Trial Therapy. Spinal cord stimulation (SCS) trial therapy activated using FDA-approved non BSC SCS system that the subject was implanted with, and received SCS therapy from, prior to study enrollment
  Interventions: Device: Non Boston Scientific SCS Trial Therapy

INTERVENTIONS:
Device: Non Boston Scientific SCS Trial Therapy — No procedures will be attempted as part of this study. This intervention refers to connection and activation of a previously implanted and programmed FDA-approved non Boston Scientific SCS trial system for 30 minutes of SCS therapy for pain
  Arms: Non Boston Scientific SCS Trial Therapy
Device: BSC approved SCS Trial Therapy w/ OMG — No procedures will be attempted as part of this study. This intervention refers to connection and activation of all Boston Scientific commercially approved SCS trial systems for 30 minutes of SCS therapy for pain
  Arms: BSC approved SCS Trial Therapy w/ OMG

SUMMARY:
The purpose of this study is to evaluate patient preference of the Boston Scientific Corporation (BSC) commercially approved spinal cord stimulation (SCS) systems with the Observational Mechanical Gateway (OMG) in patients who failed non-BSC SCS trial therapy.

DETAILED DESCRIPTION:
Spinal cord stimulation (SCS) is an established therapy for the treatment of chronic pain of the trunk and/or limbs. Standard practice includes a screening trial, typically lasting from 3 days to 7 days or more, for both the physician and the patient to evaluate whether SCS therapy is appropriate for permanent implantation. Screening trial success (hereafter referred to as a trial) is often considered predictive of long-term success of the therapy, although that has never been definitively demonstrated.

Boston Scientific Corporation (BSC) developed the Observational Mechanical Gateway (OMG) connectors to allow patients who previously underwent an SCS trial using Medtronic or St Jude Medical leads, operating room cables (OR-cables), and external trial stimulators (ETSs), to be able to connect to BSC commercially approved Spinal Cord Stimulation (SCS) trial systems to evaluate the BSC SCS therapy in the physician office setting prior to removal of the non-BSC leads.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic intractable pain of the trunk and/or lower extremities
* History of trunk and/or lower extremity pain lasting at least 6 months
* Study candidate completed a spinal cord stimulation (SCS) trial of a FDA-approved non-Boston Scientific Corporation (non-BSC) system, exclusively for the treatment of chronic intractable pain of the trunk and/or lower extremities, that will not proceed to permanent implantation due to unsatisfactory treatment or in the physician's opinion received sub-optimal results
* Currently implanted with FDA-approved non-BSC SCS lead(s) exclusively in the thoracolumbar epidural space that are temporarily anchored for non-surgical removal at the termination of the screening trial period and which are approved for use with either the Observational Mechanical Gateway (OMG) A or OMG-M, per the OMG directions for use

Key Exclusion Criteria:

* Primary source of pain is cancer-related, pelvic, visceral or angina
* Investigator-suspected gross lead migration during the non-BSC trial period which may preclude the study candidate from receiving adequate SCS therapy
* Study candidate reports <10% paresthesia coverage of overall pain while running the preferred stimulation settings on the non-BSC SCS system at the end of the non-BSC SCS screening trial period
* Study candidate unwilling to tolerate implantation with an SCS system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Corporation
Locations (13):
- United States (13):
  - Hope Research Institute, Phoenix, Arizona
  - Neurovations, Napa, California
  - Comprehensive Pain Specialists, Broomfield, Colorado
  - Coastal Orthopedics and Sports Medicine of Southwest Florida, PA, Bradenton, Florida
  - Southeastern Integrated Medical, Gainesville, Florida
  - Compass Research, LLC, Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Global Scientific Innovations - Advanced Pain Care Clinic, Evansville, Indiana
  - Columbia Interventional Pain Center, Columbia, Missouri
  - Southern New York NeuroSurgical Group, Johnson City, New York
  - New York Spine and Wellness Center, North Syracuse, New York
  - Riverhills Healthcare Incorporated, Cincinnati, Ohio
  - West Virginia University Hospitals, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment to Control: Treatment (BSC SCS Therapy) followed by Control (non-BSC SCS Therapy)
- Control to Treatment: Control (non-BSC SCS Therapy) followed by Treatment (BSC SCS Therapy)
Period: Overall Study
Arm/Group | Treatment to Control | Control to Treatment
Started | 13 | 14
Completed | 12 | 14
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment to Control | Control to Treatment | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.71) | 56 (12.02) | 56.9 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 6 | 11 | 17
Region of Enrollment: United States [Number; unit: participants] | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Subject's Treatment Preference
Description: Subject were asked if he/she prefers their current period SCS therapy over the SCS therapy he/she received during the SCS trial period prior to Baseline
Time Frame: 30 minutes after activation of stimulation
Measure: Number; unit: participants
Arm/Group | Treatment to Control | Control to Treatment
Number analyzed (Participants) | 12 | 13
participants
  Period 1 Yes, Period 2 Yes | 6 | 3
  Period 1 Yes, Period 2 No | 1 | 2
  Period 1 No, Period 2 Yes | 1 | 4
  Period 1 No, Period 2 No | 4 | 4

ADVERSE EVENTS:
Time Frame: 180 days post randomization
Arm/Group | Treatment to Control | Control to Treatment
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No